CLINICAL TRIAL: NCT07223996
Title: Use of In-Home Non-Stress Monitoring Device for Fetal Monitoring: A Nonsignificant Risk (NSR) Device Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nestmedic Spolka Akcyjna (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 004
Record Dates: First submitted 2025-10-24; First posted 2025-11-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy; Fetal Monitoring
Keywords: fetal heart rate monitoring; non-stress test; prenatal care; telemedicine; maternal health; home monitoring; PregnaOne System

STUDY DESIGN:
Intervention Model Description: Participants will complete one study visit including two monitoring sessions: (1) simultaneous use of the PregnaOne System and INVU system, and (2) self-monitoring using only the PregnaOne System. No randomization or parallel assignment is applied.
Masking Description: Open-label study. Participants and study personnel are aware of the device being used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- PregnaOne System (Experimental): Participants will use the PregnaOne System for fetal monitoring during a single study visit. Each participant will complete two monitoring sessions:
  1. Simultaneous use of the PregnaOne System and the INVU system.
  2. Self-monitoring using only the PregnaOne System. The study aims to evaluate the usability, safety, and performance of the PregnaOne System for non-stress fetal monitoring in a home-like setting.
  Interventions: Device: PregnaOne System

INTERVENTIONS:
Device: PregnaOne System — The PregnaOne System is a non-significant risk (NSR) investigational medical device designed for in-home fetal monitoring. It includes the Pregnabit Pro device and the cloud-based PregnaOne Platform software. The system records fetal heart rate, maternal pulse, and uterine activity, transmitting data to a remote monitoring center for clinical evaluation.
  During the study, participants will perform two monitoring sessions:
  1. Simultaneous use of the PregnaOne and INVU systems.
  2. Independent monitoring using only the PregnaOne System. The study evaluates the usability, safety, and performance of the PregnaOne System in comparison with a reference device.
  Other Names: Pregnabit Pro; PregnaOne Platform

SUMMARY:
This study evaluates the safety and performance of the PregnaOne System, a non-significant risk (NSR) investigational medical device for in-home fetal monitoring in pregnant women during the third trimester. The PregnaOne System consists of the Pregnabit Pro device and related software, designed to record fetal heart rate, maternal pulse, and uterine contractions in a home-like environment. The study compares the performance of the PregnaOne System with a similar FDA-cleared at-home monitoring system (the INVU system by Nuvo). Approximately 70 pregnant women will participate at three medical centers in the United States. Each participant will complete one training session and two fetal monitoring sessions during a single study visit.

DETAILED DESCRIPTION:
This is a prospective, single-visit, non-randomized, comparative study designed to evaluate the PregnaOne System, an investigational Class II medical device intended for in-home fetal monitoring. The system includes the Pregnabit Pro device and associated software that collect and transmit data on fetal heart rate, fetal movement, maternal pulse rate, and uterine muscle activity for remote review by healthcare professionals.

The goal of this study is to assess the safety, usability, and signal performance of the PregnaOne System compared to the INVU system, an FDA-cleared home fetal monitoring device. The study will be conducted under a non-significant risk (NSR) designation.

Approximately 70 pregnant women in their third trimester will be enrolled at three U.S. medical centers. Each participant will attend one in-clinic visit simulating an at-home environment. The study visit includes:

Training session - participants are instructed on how to use the PregnaOne System.

First monitoring session - a 30-minute fetal monitoring period using both the PregnaOne System and the INVU system simultaneously.

Second monitoring session - a 30-minute self-conducted monitoring session using only the PregnaOne System without staff assistance.

During each session, participants remain in a seated or reclined position and record fetal movements. Study staff will be available to assist and ensure participant safety.

No known risks are associated with fetal heart rate monitoring, though mild discomfort from device straps may occur.

Participants receive compensation for their time and travel. Study data will support the submission of a 510(k) premarket notification to the U.S. Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Able to independently read and understand written and spoken English and willing to provide written informed consent and comply with all instructions required by the study protocol.
* Female aged 22 years or older.
* Estimated gestational age between 32 and 41 weeks.
* Singleton gestation.
* Pre-pregnancy or first prenatal visit BMI < 40 kg/m².
* Able and willing to undergo fetal monitoring sessions in a simulated home environment at the study site.
* Women who do not meet the gestational age criterion at the screening visit but will meet it by the study visit (within two weeks) may be enrolled.

Exclusion Criteria:

* In active labor or in the delivery room during labor.
* Requires hospitalization or life support.
* Any contraindications for cardiotocography (CTG) monitoring.
* Severe hypertension (≥160/110 mmHg measured twice, 15 minutes apart).
* Known allergy to latex, ultrasound (US) gel, or ECG gel.
* Skin conditions (e.g., edema, erythema, irritation, infection, lesions, or open wounds) at contact points for the Pregnabit Pro or comparator devices.
* Implanted electronic devices (e.g., pacemaker, stimulator, defibrillator, pump).
* Members of vulnerable populations other than pregnant women (e.g., minors, wards of the state, cognitively impaired individuals, prisoners, or institutionalized persons).

Min Age: 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Agreement Between PregnaOne System and Comparator Device (INVU System) for Fetal Heart Rate (fHR) Measurements | At single study visit (Day 1)
  To assess the agreement between fetal heart rate (fHR) measurements obtained with the PregnaOne System and those obtained with the comparator device during simultaneous monitoring. Agreement will be evaluated using correlation and Bland-Altman analysis.
Agreement Between PregnaOne System and Comparator Device (INVU System) for Uterine Muscle Activity Measurements | At single study visit (Day 1)
  To assess the agreement between uterine muscle activity measurements obtained with the PregnaOne System and those obtained with the comparator device during simultaneous monitoring. Agreement will be evaluated using correlation and Bland-Altman analysis.
Percent of Participants Who Obtain a Quality Maternal Pulse Rate (mPR) Recording | At single study visit (Day 1)
  To determine the proportion of participants who obtain a quality maternal pulse rate (mPR) recording during simultaneous monitoring, defined as a valid and stable signal without major artifacts.
Percent of Participants Who Successfully Complete a Self-Monitoring Session | At single study visit (Day 1)
  To assess the ability of participants to successfully complete a self-monitoring session in a simulated home environment, including correct device placement and successful recording of signals, as determined by a healthcare professional (HCP).
Agreement Between PregnaOne System and Comparator for Fetal Heart Rate (fHR) | At single study visit (Day 1)
  To evaluate the agreement between fetal heart rate (fHR) measurements obtained using the PregnaOne System and those obtained using the comparator device. fHR data will be analyzed to determine correlation, limits of agreement, and measurement bias between the two systems.
Agreement Between PregnaOne System and Comparator for Uterine Muscle Activity | At single study visit (Day 1)
  To evaluate the agreement between uterine muscle activity measurements obtained using the PregnaOne System and those obtained using the comparator device. Data will be analyzed to determine correlation, limits of agreement, and measurement bias.

SECONDARY OUTCOMES:
Percent of Participants Who Obtain a Quality Maternal Pulse Rate (mPR) Recording | At single study visit (Day 1)
  To determine the percentage of participants who obtain a quality mPR recording during simultaneous monitoring using the PregnaOne System.
Percent of Participants Who Successfully Place the Device | At single study visit (Day 1)
  To determine the percentage of participants who successfully place the PregnaOne device as determined by a healthcare professional (HCP) during self-monitoring.
Percent of Participants Who Obtain a Quality Recording of fHR, Uterine Muscle Activity, and mPR During Self-Monitoring | At single study visit (Day 1)
  To determine the percentage of participants who obtain a quality recording of fetal heart rate (fHR), uterine muscle activity, and maternal pulse rate (mPR) during self-monitoring, as assessed by a healthcare professional (HCP).

OTHER OUTCOMES:
Frequency, Type, and Severity of Adverse Events (AEs) and Adverse Device Effects (ADEs) | Throughout the study duration (up to 1 day per participant)
  To assess the safety and tolerability of the PregnaOne System when used in pregnant women 32-41 weeks of gestation. The frequency, types, and severities of adverse events (AEs) and adverse device effects (ADEs), and their relationship to the devices or study procedures, will be summarized descriptively for both the PregnaOne System and the comparator. This endpoint is descriptive only and includes data from both Stage 1 (Simultaneous Monitoring) and Stage 2 (Self-Monitoring).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Szopa, Study Director — Nestmedic Spolka Akcyjna; Jacek Gnich, Study Chair — Nestmedic Spolka Akcyjna
Locations (3):
- United States (3):
  - Christie Clinic, LLC, Champaign, Illinois
  - The Iowa Clinic, P.C., West Des Moines, Iowa
  - Wilmington Health, PLLC, Wilmington, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Official website of Nestmedic S.A., the sponsor of the study. — http://nestmedic.com
- See also: Official website of the Pregnabit® system, a telemedical solution for remote fetal monitoring. — http://pregnabit.com